CLINICAL TRIAL: NCT05016375
Title: An Exploration of People's Perceptions of Undertaking Passive Heating as a Treatment for Type 2 Diabetes Mellitus
Brief Title: Perceptions of Passive Heating in Individuals With T2DM
Status: Completed | Type: Observational
Sponsor: University of Portsmouth (Other)
Collaborators: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Principal Investigator, Ant Shepherd, Senior lecturer, University of Portsmouth
Other Study IDs: 008AS
Record Dates: First submitted 2021-07-20; First posted 2021-08-23 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes
Keywords: Passive heating
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- T2DM: Individuals with T2DM.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Interview with individuals with T2DM

SUMMARY:
Current treatments for type 2 diabetes (e.g., lifestyle changes and clinical interventions such as medication), have been shown to be unsustainable due to low levels of physical activity and increasing clinical costs. Therefore, scientists have been looking for new treatments to address this issue. One such treatment that is being investigated is passive heating (e.g., hot baths, saunas, etc.). In this study the investigators want to ascertain what passive heating, if any, individuals with T2DM currently do, what their perceptions of passive heating would be if it were to become a treatment, what may make it easier or more difficult for them to engage in passive heating, and how this might impact other areas of their life such as physical activity.

DETAILED DESCRIPTION:
This study employs an interpretivist approach through semi-structured interviews to highlight participants' perceptions of and experiences with passive heating. To date, this topic has not been explored in-depth - this approach should bring nuance and context to light, aiding in future advocacy work which explores the potential of passive heating as a viable treatment for adults with T2DM.

Semi-structured interviews will be facilitated by an interview guide consisting of four main topic areas aiming to explore an individual's perception of and experience with passive heating as a treatment for T2DM and to ascertain whether engaging in this behaviour may affect physical activity. As no two conversations are ever the same, the approach to the interviews is one of flexibility through the use of open-ended questions and potential probes as the situation dictates - remaining open to following particular lines of participant thought.

Interviews will all be conducted by the Principal investigator, Mr Thomas James, a doctoral researcher who has been trained in the required skills. He has also undertaken necessary training in Good Clinical Practice and Valid Informed Consent. Interviews will be conducted virtually, by telephone or in person and will take place either at home or in a laboratory setting, dependent upon the individual's wishes. The interviews will be audio recorded and subsequently transcribed verbatim by a member of the research team. Transcriptions will be analysed via thematic analysis to determine the main themes expressed by participants. All data analysis will be conducted by a trained member of the research team.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Willing and able to undertake the interview process
* Able to give informed consent

Exclusion Criteria:

* Age < 18 years
* Does not provide written informed consent
* Any neurological/psychiatric diagnoses
* Lack of fluency in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with T2DM
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Explore bathing and spa behaviour by applying the social-ecological model to interpretivist thematic analysis. | ~1 hour interview
  To explore the current bathing and spa behaviours among individuals living with T2DM and their perceptions regarding passive heating as a treatment.

SECONDARY OUTCOMES:
Explore perceived facilitators and barriers to passive heating by applying the social-ecological model to interpretivist thematic analysis. | ~1 hour interview
  To explore how participants perceive as the facilitators and barriers to engaging in passive heating within and outside the home.
Explore how passive heating might impact physical activity by applying the social-ecological model to interpretivist thematic analysis. | ~1 hour interview
  To explore how engaging in passive heating might impact the physical activity of individuals with T2DM.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sport and Exercise Science, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No